CLINICAL TRIAL: NCT04881448
Title: Evaluation of Homogeneity Between eGFR Slopes Derived From Retrospective Clinical Practice Data and eGFR Slopes Derived From Prospectively Collected, Protocol-driven Data
Brief Title: A Study to Examine Past Estimated Glomerular Filtration Rate (eGFR) Slope as a Risk Marker for Rapid Kidney Function Decline in People With Chronic Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1366-0026
Record Dates: First submitted 2021-05-04; First posted 2021-05-11 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with chronic kidney disease - overall population (Experimental): Patients with chronic kidney disease (CKD), including patients with non-diabetic chronic kidney disease (non-DKD) and diabetic kidney disease (DKD). Participants in this study did not receive any medication or study drug.
  Interventions: Diagnostic Test: collection of serum/capillary creatinine values

INTERVENTIONS:
Diagnostic Test: collection of serum/capillary creatinine values — collection of serum/capillary creatinine values

SUMMARY:
This study is intended to investigate the usefulness of estimated glomerular filtration rate (eGFR) slopes derived from retrospective routine clinical practice data, compare those retrospective slopes with those generated in a prospective fashion and successively identify rapidly progressing chronic kidney disease (CKD) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent in accordance with International Council on Harmonisation - Good Manufacturing Practice (ICH-GCP) and local legislation prior to admission to the trial.
2. Patients with available medical records for data abstraction to meet the objectives of the study.
3. Male or female patients aged ≥ 18 years at time of consent.
4. Body Mass Index (BMI) ≥ 18.5 and < 50 kg/m² at Visit 1.
5. Clinical diagnosis of Chronic Kidney Disease (CKD).
6. Estimated Glomerular Filtration Rate (eGFR) decline of at least 1ml/min/1.73m²/year based on historical data from (electronic) medical records.
7. eGFR (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) 20 - 90 ml/min/1.73m² at Visit 1 calculated from serum creatinine measured by a central laboratory.
8. Patients are expected to be on optimal and stable background treatment (according to local therapy guidelines).
9. At least 4 serum creatinine values in the retrospective phase:

   * The most recent creatinine value not more than 6 months prior to Visit 1 (Screening Visit).
   * The most recent and oldest serum creatinine values should be no less than 1 year apart and no greater than 5 years apart.
   * There should be no gap of creatinine values of 2 years or longer.

Exclusion Criteria:

1. Changes in CKD or other key background treatments (including dose changes) known to impact eGFR values, over the past 4 weeks for Angiotensin Converting Enzyme inhibitors (ACEis) and Angiotensin Receptor Blockers (ARBs) and 8 weeks for Sodium-Glucose Co-Transporter-2 (SGLT2) inhibitors prior to Screening.
2. Autosomal Dominant Polycystic Kidney Disease (ADPKD), uncontrolled lupus nephritis, in the opinion of investigators.
3. Any iv immune suppression therapy within the last 3 months prior to Visit 1 or anyone currently on >45 mg prednisolone (or equivalent).
4. Acute kidney injury (AKI) according to the Kidney Disease: Improving Global Outcomes (KDIGO) definition in the 30 days prior to Visit 1 until the start of trial assessments.
5. Planned start of chronic renal replacement therapy during the trial or end stage renal disease (i.e < 15 ml/min at 2 measurements 30 days apart) before start of trial assessments.
6. Medical history of cancer or treatment for cancer in the last two years prior to Visit 1 (except appropriately treated basal cell carcinoma of the skin, in situ carcinoma of uterine cervix, and prostatic cancer of low grade [T1 or T2]).
7. Major surgery (investigator's judgement) planned during the trial.
8. Currently enrolled in an investigational device or drug trial, i.e., less than 30 days before Visit 1 since ending an investigational device or drug trial(s) or receiving investigational treatment(s).

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (19):
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - Desert Cities Dialysis - Amethyst, Victorville, California
  - Kidney & Hypertension Center, Victorville, California
  - Davita Clinical Research-Hartford, Bloomfield, Connecticut
  - Nephrology & Hypertension Assoc., PC, Middlebury, Connecticut
  - Med-Care Research, Miami, Florida
  - International Research Associates, Miami, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - DaVita Clinical Research, Edina, Minnesota
  - DaVita Clinical Research, Las Vegas, Nevada
  - Kidney Medical Associates, PLLC, The Bronx, New York
  - DaVita Clinical Research (DCR) Spartanburg, Spartanburg, South Carolina
  - Davita Clinical Research, El Paso, Texas
  - Sunbeam Clinical Research, Greenville, Texas
  - DaVita Clinical Research, Houston, Texas
  - DaVita Clinical Research, San Antonio, Texas
  - DaVita Clinical Research, The Woodlands, Texas
  - Tidewater Kidney Specialists, Chesapeake, Virginia
  - DaVita Clinical Research, Wauwatosa, Wisconsin
- Germany (3):
  - DaVita Clinical Research Germany GmbH, Düsseldorf
  - InnoDiab Forschung GmbH, Essen
  - DaVita Clinical Research Germany GmbH, Geilenkirchen
- Hungary (2):
  - DRC Drug Research Ltd, Balatonfüred
  - Szent Imre Korhaz, Budapest, Budapest
- Hospital Virgen Macarena, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicentre, non-randomised, low-intervention study that did not involve administration of study drug, which aimed to investigate the estimated Glomerular Filtration Rate (eGRF) slopes derived from retrospective routine clinical practice data, compare those retrospective slopes with those generated in a prospective fashion and successively identify rapidly progressing chronic kidney disease (CKD) patients.
Pre-assignment Details: Patients were screened for eligibility prior to participation in the trial. They underwent a screening period of up to 2 weeks from the time of informed consent. Patients who successfully completed the screening and met all inclusion criteria, including the availability of requisite historical eGFR data, and did not meet any of the exclusion criteria, qualified for enrolment into the 48 weeks prospective phase of the study.
Groups:
- Patients With Chronic Kidney Disease - Overall Population: Patients with chronic kidney disease (CKD), including patients with non-diabetic chronic kidney disease (non-DKD) and diabetic chronic kidney disease (DKD). This study did not involve administration of study drug.
Period: Overall Study
Arm/Group | Patients With Chronic Kidney Disease - Overall Population
Started | 223
Completed | 0
Not Completed | 223
Not completed — Study cancelled by sponsor | 220
Not completed — Withdrawal by Subject | 2
Not completed — Exhausted all attempts to contact subject | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): FAS includes all patients entered into the 48-week prospective phase of the study who have at least one post-baseline assessment.
Arm/Group | Patients With Chronic Kidney Disease - Overall Population
Number analyzed (Participants) | 210
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 190
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 46
  White | 150
  More than one race | 1
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Homogeneity (eGFR Slope Shift Table) Between eGFR Slopes Derived From Retrospective and Prospective eGFR Values
Description: Retrospective and prospective slopes were derived using a linear random slope model. The prospective estimated Glomerular Filtration Rate (eGFR) slope for each patient was derived using eGFR values in the prospective phase as the dependent variable and time in the prospective phase as the continuous independent variable with random intercept and random slope. The retrospective eGFR slope for each patient was derived similarly using the data in the retrospective phase, and the time in the retrospective phase calculated relative to the first retrospective measurement per patient.
  Homogeneity was primarily evaluated via a shift analysis with categories of eGFR decline rate of 1 to < 3 (slow) and >= 3 ml/min/1.73m2/year (fast), in each of the retrospective and prospective phases.
  eGFR data collected 4 weeks before acute kidney injury and up to 8 weeks after acute kidney injury, and eGFR data occurring after changes to baseline background therapy (SGLT2i/ACEi/ARB) were excluded.
Time Frame: Prospective slopes: All measurements from baseline until the last available visit were considered for inclusion in the estimation, including unscheduled visits, up to 48 weeks. Retrospective slopes: up to 66 months.
Population: Full Analysis Set (FAS): FAS includes all patients entered into the 48-week prospective phase of the study who have at least one post-baseline assessment. Summary statistics are reported by overall and DKD/non-DKD patient populations. The n's in each category for DKD/non-DKD may not add up to the overall number, since separate random slope models are used leading to differences in estimated eGFR slope in each of the calculations.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Diabetic Chronic Kidney Disease - Patient Population: Patients with diabetic chronic kidney disease (DKD).
- Patients With Non-diabetic Chronic Kidney Disease - Patient Population: Patients with non-diabetic chronic kidney disease (non-DKD).
Arm/Group | Patients With Diabetic Chronic Kidney Disease - Patient Population | Patients With Non-diabetic Chronic Kidney Disease - Patient Population | Patients With Chronic Kidney Disease - Overall Population
Number analyzed (Participants) | 114 | 96 | 210
Participants
  Retrospective Phase: > -1 | 9 | 15 | 21
  Retrospective Phase: > -3 to -1 | 27 | 20 | 43
  Retrospective Phase: <= -3 | 78 | 61 | 146
  from > -1 (in Retrospective Phase) to > -1 (in Prospective Phase): number analyzed (Participants) | 9 | 15 | 21
  from > -1 (in Retrospective Phase) to > -1 (in Prospective Phase) | 4 | 8 | 9
  from > -1 (in Retrospective Phase) to > -3 to -1 (in Prospective Phase): number analyzed (Participants) | 9 | 15 | 21
  from > -1 (in Retrospective Phase) to > -3 to -1 (in Prospective Phase) | 1 | 1 | 2
  from > -1 (in Retrospective Phase) to <= -3 (in Prospective Phase): number analyzed (Participants) | 9 | 15 | 21
  from > -1 (in Retrospective Phase) to <= -3 (in Prospective Phase) | 4 | 6 | 10
  from > -3 to -1 (in Retrospective Phase) to > -1 (in Prospective Phase): number analyzed (Participants) | 27 | 20 | 43
  from > -3 to -1 (in Retrospective Phase) to > -1 (in Prospective Phase) | 12 | 7 | 18
  from > -3 to -1 (in Retrospective Phase) to > -3 to -1 (in Prospective Phase): number analyzed (Participants) | 27 | 20 | 43
  from > -3 to -1 (in Retrospective Phase) to > -3 to -1 (in Prospective Phase) | 6 | 2 | 5
  from > -3 to -1 (in Retrospective Phase) to <= -3 (in Prospective Phase): number analyzed (Participants) | 27 | 20 | 43
  from > -3 to -1 (in Retrospective Phase) to <= -3 (in Prospective Phase) | 9 | 11 | 20
  from <= -3 (in Retrospective Phase) to > -1 (in Prospective Phase): number analyzed (Participants) | 78 | 61 | 146
  from <= -3 (in Retrospective Phase) to > -1 (in Prospective Phase) | 45 | 6 | 39
  from <= -3 (in Retrospective Phase) to > -3 to -1 (in Prospective Phase): number analyzed (Participants) | 78 | 61 | 146
  from <= -3 (in Retrospective Phase) to > -3 to -1 (in Prospective Phase) | 11 | 3 | 41
  from <= -3 (in Retrospective Phase) to <= -3 (in Prospective Phase): number analyzed (Participants) | 78 | 61 | 146
  from <= -3 (in Retrospective Phase) to <= -3 (in Prospective Phase) | 22 | 52 | 66

ADVERSE EVENTS:
Time Frame: From signing the informed consent onwards until the end of study visit, up to 50 weeks.
Description: Full Analysis Set (FAS): FAS includes all patients entered into the 48-week prospective phase of the study who have at least one post-baseline assessment.
Arm/Group | Patients With Chronic Kidney Disease - Overall Population
All-Cause Mortality (participants affected / at risk) | 0/210
Serious Adverse Events (participants affected / at risk) | 0/210
Other Adverse Events (participants affected / at risk) | 0/210

LIMITATIONS AND CAVEATS:
The study was terminated prematurely, due to decision of the sponsor. Due to the early study termination leading to a short follow up time and limited number of eGFR assessments in the prospective phase, the results need to be interpreted cautiously.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT04881448/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04881448/SAP_001.pdf